CLINICAL TRIAL: NCT04761198
Title: A Phase 1b/2 Open-Label Study of the Efficacy and Safety of Etigilimab (MPH313) Administered in Combination With Nivolumab to Subjects With Locally Advanced or Metastatic Solid Tumors (ACTIVATE)
Brief Title: A Study of Etigilimab and Nivolumab in Participants With Locally Advanced or Metastatic Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mereo BioPharma (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MPH313-1-02; 2020-004222-37 (EudraCT Number)
Record Dates: First submitted 2021-02-12; First posted 2021-02-18 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumor, Adult; Advanced Solid Tumor; Metastatic Solid Tumor
Keywords: etigilimab; nivolumab; anti-TIGIT antibody; MPH313; Opdivo; ACTIVATE
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Basket study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort A: Endometrial Cancer CPI (PD-1/PD-L1) Naive (Experimental): Participants with endometrial cancer CPI (programmed death-1 [PD-1]/ programmed death ligand-1 [PD-L1]) naive will receive etigilimab in combination with nivolumab every 2 weeks and will continue treatment until protocol-defined discontinuation criteria are met.
  Interventions: Drug: Etigilimab; Drug: Nivolumab
- Cohort B: Head and Neck Squamous Cell Carcinoma (Experimental): Participants with head and neck cell carcinoma will receive etigilimab in combination with nivolumab every 2 weeks and will continue treatment until protocol-defined discontinuation criteria are met.
  Interventions: Drug: Etigilimab; Drug: Nivolumab
- Cohort C: Cervical Carcinoma (Experimental): Participants with cervical carcinoma will receive etigilimab in combination with nivolumab every 2 weeks and will continue treatment until protocol-defined discontinuation criteria are met.
  Interventions: Drug: Etigilimab; Drug: Nivolumab
- Cohort D (Recurrent Advanced and/or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma) (Experimental): Participants with recurrent advanced and/or metastatic gastric or gastroesophageal junction adenocarcinoma will receive etigilimab in combination with nivolumab every 2 weeks and will continue treatment until protocol-defined discontinuation criteria are met.
  Interventions: Drug: Etigilimab; Drug: Nivolumab
- Cohort E: TMB-H + MSS Solid Tumors (Experimental): Participants with tumour mutational burden-high (TMB-H) and microsatellite stable (MSS) solid tumors will receive etigilimab in combination with nivolumab every 2 weeks and will continue treatment until protocol-defined discontinuation criteria are met.
  Interventions: Drug: Etigilimab; Drug: Nivolumab
- Cohort F: Rare Tumors (Sarcoma, Uveal Melanoma, Germ Cell) (Experimental): Participants with rare tumors (sarcoma, uveal melanoma, and germ cell) will receive etigilimab in combination with nivolumab every 2 weeks and will continue treatment until protocol-defined discontinuation criteria are met.
  Interventions: Drug: Etigilimab; Drug: Nivolumab
- Cohort G: Endometrial Cancer Post- CPI (PD-1/PD-L1 Treated) (Experimental): Participants with endometrial cancer (PD-1/PD-L1 treated) will receive etigilimab in combination with nivolumab every 2 weeks and will continue treatment until protocol-defined discontinuation criteria are met.
  Interventions: Drug: Etigilimab; Drug: Nivolumab
- Cohort H: Ovarian Cancer (Experimental): Participants with ovarian cancer will receive etigilimab in combination with nivolumab every 2 weeks and will continue treatment until protocol-defined discontinuation criteria are met.
  Interventions: Drug: Etigilimab; Drug: Nivolumab

INTERVENTIONS:
Drug: Etigilimab — IV infusion of IV etigilimab every 2 weeks
  Other Names: MPH313
Drug: Nivolumab — IV infusion of nivolumab every 2 weeks
  Other Names: Opdivo

SUMMARY:
This is an open-label, phase 1b/2, multicenter study designed to evaluate the efficacy, safety, tolerability, pharmacokinetics (PK), and pharmacodynamics of etigilimab in combination with nivolumab in participants with locally advanced or metastatic solid tumors. Participants will be assigned to receive etigilimab (every 2 weeks) in combination with nivolumab (240 milligrams [mg] every 2 weeks).

DETAILED DESCRIPTION:
This is an open-label, phase 1b/2, multicenter study designed to evaluate the efficacy, safety, tolerability, PK, and pharmacodynamics of etigilimab in combination with nivolumab in participants with locally advanced or metastatic solid tumors. Participants will be assigned to receive etigilimab (every 2 weeks) in combination with nivolumab (240 mg every 2 weeks) and will continue until either unacceptable toxicity or disease progression. Participants may continue to receive treatment beyond documented Response Evaluation Criteria in Solid Tumours Version 1.1 (RECIST v1.1) or disease progression. Participants who are both checkpoint inhibitor (CPI) naive as well as participants who have received or progressed following a CPI will be eligible and include the following tumor types: head and neck squamous cell carcinoma (HNSCC), cervical carcinoma, gastric or gastroesophageal carcinoma, endometrial carcinoma, tumor mutation burden high (TMB-H), select rare tumors and ovarian carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of a relevant tumor type as per the study protocol and not candidates for curative surgery or radiation therapy
* Available tumor tissue (archival or newly obtained core or excisional biopsy)
* Adequate hematologic and end organ function as measured by laboratory screening panel in the 14 days prior to treatment
* Life expectancy greater than 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Adequate contraception for women of childbearing potential
* Pre-specified wash-out of prior anti-PD1/PDL-1 therapy

Exclusion Criteria:

* Concurrent active malignancy
* Major surgery within 4 weeks of treatment
* Participants with active, known or suspected autoimmune diseases
* Prior treatment with cluster of differentiation (CD) 137 agonists, anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) and anti-T-cell immunoreceptor with immunoglobulin (Ig) and immunoreceptor tyrosine-based inhibitory motif domains (TIGIT) antibodies
* History of any Grade 3 or 4 immune-related adverse event (AE) toxicity from prior immunotherapy that resulted in treatment discontinuation
* History of immune-related adverse events that lead to discontinuation of anti-PD-1 or PDL-1 therapy
* Active infections of human immunodeficiency virus (HIV), hepatitis B, hepatitis C
* Medical illness or abnormal laboratory finding that would, in the Study Investigator's judgement, increase the risk to the participant associated with participation in the study
* Pregnancy in female participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (14):
  - Mereo Investigator Site, Phoenix, Arizona
  - Mereo Investigator Site, Greenbrae, California
  - Mereo Investigator Site, Los Angeles, California
  - Mereo Investigator Site, Jacksonville, Florida
  - Mereo Investigator Site, Boston, Massachusetts
  - Mereo Investigator Site, Ann Arbor, Michigan
  - Mereo Investigator Site, Rochester, Minnesota
  - Mereo Investigator Site, New York, New York
  - Mereo Investigator Site, Durham, North Carolina
  - Mereo Investigator Site, Oklahoma City, Oklahoma
  - Mereo Investigator Site, Nashville, Tennessee
  - Mereo Investigator Site, Houston, Texas
  - Mereo Investigator Site, West Valley City, Utah
  - Mereo Investigator Site, Fairfax, Virginia
- United Kingdom (2):
  - Royal Marsden, London
  - Sarah Cannon UK, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Cohort D (Recurrent advanced and/or metastatic gastric or gastroesophageal junction adenocarcinoma) did not enroll any participants due to closure of the cohort by the Sponsor.
Groups:
- Cohort A: Endometrial Cancer CPI (PD-1/PD-L1) Naive: Participants with endometrial cancer checkpoint inhibitors (CPI) (programmed death-1 [PD-1]/ programmed death ligand-1 [PD-L1]) naive received etigilimab in combination with nivolumab every 2 weeks and continued treatment until protocol-defined discontinuation criteria were met.
- Cohort B: Head and Neck Squamous Cell Carcinoma: Participants with head and neck cell carcinoma received etigilimab in combination with nivolumab every 2 weeks and continued treatment until protocol-defined discontinuation criteria were met.
- Cohort C: Cervical Carcinoma: Participants with cervical carcinoma received etigilimab in combination with nivolumab every 2 weeks and continued treatment until protocol-defined discontinuation criteria were met.
- Cohort E: TMB-H + MSS Solid Tumors: Participants with tumour mutational burden-high (TMB-H) and microsatellite stable (MSS) solid tumors received etigilimab in combination with nivolumab every 2 weeks and continued treatment until protocol-defined discontinuation criteria were met.
- Cohort F: Rare Tumors (Sarcoma, Uveal Melanoma, Germ Cell): Participants with rare tumors (sarcoma, uveal melanoma, and germ cell) received etigilimab in combination with nivolumab every 2 weeks and continued treatment until protocol-defined discontinuation criteria were met.
- Cohort G: Endometrial Cancer Post- CPI (PD-1/PD-L1 Treated): Participants with endometrial cancer (PD-1/PD-L1 treated) received etigilimab in combination with nivolumab every 2 weeks and continued treatment until protocol-defined discontinuation criteria were met.
- Cohort H: Ovarian Cancer: Participants with ovarian cancer received etigilimab in combination with nivolumab every 2 weeks and continued treatment until protocol-defined discontinuation criteria were met.
Period: Overall Study
Arm/Group | Cohort A: Endometrial Cancer CPI (PD-1/PD-L1) Naive | Cohort B: Head and Neck Squamous Cell Carcinoma | Cohort C: Cervical Carcinoma | Cohort E: TMB-H + MSS Solid Tumors | Cohort F: Rare Tumors (Sarcoma, Uveal Melanoma, Germ Cell) | Cohort G: Endometrial Cancer Post- CPI (PD-1/PD-L1 Treated) | Cohort H: Ovarian Cancer
Started | 11 | 1 | 8 | 9 | 33 | 4 | 10
Received at Least 1 Dose of Study Drug | 11 | 1 | 8 | 9 | 33 | 4 | 10
Response-Evaluable (RE) Analysis Set (Participants with measurable disease at baseline who received study drug and had at least 1 post-baseline response assessment or discontinued treatment due to disease progression (including death due to disease progression) within 16 weeks (+ a 2-week window) of the first dose of study drug.) | 10 | 1 | 8 | 9 | 31 | 3 | 10
Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not Completed | 11 | 1 | 8 | 9 | 32 | 4 | 10
Not completed — Progressive Disease | 1 | 0 | 0 | 1 | 4 | 1 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 2 | 1 | 2 | 5 | 14 | 2 | 5
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 0 | 2 | 0 | 1
Not completed — Study Terminated by Sponsor | 6 | 0 | 5 | 3 | 10 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received any amount of study drug.
Groups:
- Cohort A: Endometrial Cancer CPI (PD-1/PD-L1) Naive: Participants with endometrial cancer CPI (PD-1/PD-L1) naive received etigilimab in combination with nivolumab every 2 weeks and continued treatment until protocol-defined discontinuation criteria were met.
- Cohort E: TMB-H + MSS Solid Tumors: Participants with TMB-H and MSS solid tumors received etigilimab in combination with nivolumab every 2 weeks and continued treatment until protocol-defined discontinuation criteria were met.
- Total: Total of all reporting groups
Arm/Group | Cohort A: Endometrial Cancer CPI (PD-1/PD-L1) Naive | Cohort B: Head and Neck Squamous Cell Carcinoma | Cohort C: Cervical Carcinoma | Cohort E: TMB-H + MSS Solid Tumors | Cohort F: Rare Tumors (Sarcoma, Uveal Melanoma, Germ Cell) | Cohort G: Endometrial Cancer Post- CPI (PD-1/PD-L1 Treated) | Cohort H: Ovarian Cancer | Total
Number analyzed (Participants) | 11 | 1 | 8 | 9 | 33 | 4 | 10 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (10.20) | 69.0 | 49.1 (13.53) | 62.0 (10.14) | 55.8 (13.90) | 65.3 (11.79) | 68.1 (11.43) | 59.5 (13.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 0 | 8 | 4 | 10 | 4 | 10 | 47
  Male | 0 | 1 | 0 | 5 | 23 | 0 | 0 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 5
  Not Hispanic or Latino | 10 | 1 | 8 | 8 | 30 | 4 | 10 | 71
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 3
  White | 10 | 1 | 8 | 9 | 31 | 2 | 8 | 69
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) as Assessed Based on Response Evaluation Criteria in Solid Tumours Version 1.1 (RECIST v1.1)
Description: The ORR was defined as the percentage of participants who achieved a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR) per RECIST v1.1. CR: Disappearance of all target or non-target lesions and normalization of tumor marker level. Any pathological lymph node (whether target or non-target) must have reduction in short axis to <10 millimeters (mm). PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose of study drug until the date of first objective response (CR or PR) (maximum exposure: 638 days)
Population: RE Analysis Set included all participants with measurable disease at baseline who received study drug and had at least 1 post-baseline response assessment or discontinued treatment due to disease progression (including death due to disease progression) within 16 weeks (+ a 2-week window) of the first dose of study drug. Per planned analysis, the efficacy data for Cohort F were collected and analyzed separately per tumor type.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort F: Rare Tumors (Uveal): Participants with rare tumors (uveal) received etigilimab in combination with nivolumab every 2 weeks and continued treatment until protocol-defined discontinuation criteria were met.
- Cohort F: Rare Tumors (De-diff LPS): Participants with rare tumors (de-differentiated liposarcoma [de-diff LPS]) received etigilimab in combination with nivolumab every 2 weeks and continued treatment until protocol-defined discontinuation criteria were met.
- Cohort F: Rare Tumors (UPS): Participants with rare tumors (undifferentiated pleomorphic sarcoma [UPS]) received etigilimab in combination with nivolumab every 2 weeks and continued treatment until protocol-defined discontinuation criteria were met.
- Cohort F: Rare Tumors (Other Sarcoma): Participants with rare tumors (other sarcoma) received etigilimab in combination with nivolumab every 2 weeks and continued treatment until protocol-defined discontinuation criteria were met.
- Cohort F: Rare Tumors (GCT): Participants with rare tumors (germ cell tumours [GCT]) received etigilimab in combination with nivolumab every 2 weeks and continued treatment until protocol-defined discontinuation criteria were met.
Arm/Group | Cohort A: Endometrial Cancer CPI (PD-1/PD-L1) Naive | Cohort B: Head and Neck Squamous Cell Carcinoma | Cohort C: Cervical Carcinoma | Cohort E: TMB-H + MSS Solid Tumors | Cohort F: Rare Tumors (Uveal) | Cohort F: Rare Tumors (De-diff LPS) | Cohort F: Rare Tumors (UPS) | Cohort F: Rare Tumors (Other Sarcoma) | Cohort F: Rare Tumors (GCT) | Cohort G: Endometrial Cancer Post- CPI (PD-1/PD-L1 Treated) | Cohort H: Ovarian Cancer
Number analyzed (Participants) | 10 | 1 | 8 | 9 | 8 | 10 | 6 | 3 | 4 | 3 | 10
percentage of participants | 20.0 [2.52 to 55.61] | 0 [0.00 to 97.50] | 37.5 [8.52 to 75.51] | 0 [0.00 to 33.63] | 25.0 [3.19 to 65.09] | 10.0 [0.25 to 44.50] | 16.7 [0.42 to 64.12] | 0 [0.00 to 70.76] | 0 [0.00 to 60.24] | 0 [0.00 to 70.76] | 10.0 [0.25 to 44.50]

2. Secondary Outcome: Number of Participants WithTreatment-emergent Adverse Events (TEAEs), Any Adverse Events of Special Interests (AESIs), AESI Immune Related AEs, and AESI Infusion Reactions
Description: TEAEs were defined as adverse events (AEs) with an onset date on or after the date of first administration of study drug up to 100 days after the last dose of study drug and before starting any subsequent cancer treatment. An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AESIs were defined as events (serious or non-serious) which were of scientific and medical concern specific to the sponsor's product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor might be appropriate. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: From first dose of study drug until 100 days after the last dose of study drug or the initiation of any subsequent cancer treatment, whichever occurs first (maximum exposure: 638 days)
Population: Safety Analysis Set included all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Endometrial Cancer CPI (PD-1/PD-L1) Naive | Cohort B: Head and Neck Squamous Cell Carcinoma | Cohort C: Cervical Carcinoma | Cohort E: TMB-H + MSS Solid Tumors | Cohort F: Rare Tumors (Sarcoma, Uveal Melanoma, Germ Cell) | Cohort G: Endometrial Cancer Post- CPI (PD-1/PD-L1 Treated) | Cohort H: Ovarian Cancer
Number analyzed (Participants) | 11 | 1 | 8 | 9 | 33 | 4 | 10
Participants
  Any TEAEs | 11 | 1 | 8 | 8 | 33 | 4 | 9
  Any AESIs | 4 | 0 | 3 | 0 | 5 | 0 | 1
  AESI Immune Related AEs | 2 | 0 | 2 | 0 | 3 | 0 | 1
  AESI Infusion Reactions | 2 | 0 | 1 | 0 | 2 | 0 | 0

3. Secondary Outcome: Disease Control Rate (DCR) as Assessed Based on RECIST v1.1
Description: The DCR was defined as the percentage of participants who achieved CR, PR, and stable disease (SD). CR: Disappearance of all target or non-target lesions and normalization of tumor marker level. Any pathological lymph node (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. SD: Persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits; and no new lesions.
Time Frame: From first dose of study drug until the date of first BOR (CR, PR, or SD) (maximum exposure: 638 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort F: Rare Tumors (De-diff LPS): Participants with rare tumors (de-diff LPS) received etigilimab in combination with nivolumab every 2 weeks and continued treatment until protocol-defined discontinuation criteria were met.
- Cohort F: Rare Tumors (UPS): Participants with rare tumors (UPS) received etigilimab in combination with nivolumab every 2 weeks and continued treatment until protocol-defined discontinuation criteria were met.
- Cohort F: Rare Tumors (GCT): Participants with rare tumors (GCT) received etigilimab in combination with nivolumab every 2 weeks and continued treatment until protocol-defined discontinuation criteria were met.
Arm/Group | Cohort A: Endometrial Cancer CPI (PD-1/PD-L1) Naive | Cohort B: Head and Neck Squamous Cell Carcinoma | Cohort C: Cervical Carcinoma | Cohort E: TMB-H + MSS Solid Tumors | Cohort F: Rare Tumors (Uveal) | Cohort F: Rare Tumors (De-diff LPS) | Cohort F: Rare Tumors (UPS) | Cohort F: Rare Tumors (Other Sarcoma) | Cohort F: Rare Tumors (GCT) | Cohort G: Endometrial Cancer Post- CPI (PD-1/PD-L1 Treated) | Cohort H: Ovarian Cancer
Number analyzed (Participants) | 10 | 1 | 8 | 9 | 8 | 10 | 6 | 3 | 4 | 3 | 10
percentage of participants | 50.0 [18.71 to 81.29] | 0 [0.00 to 97.50] | 62.5 [24.49 to 91.48] | 33.3 [7.49 to 70.07] | 50.0 [15.70 to 84.3] | 50.0 [18.71 to 81.29] | 33.3 [4.33 to 77.72] | 33.3 [0.84 to 90.57] | 0 [0.00 to 60.24] | 0 [0.00 to 70.76] | 60.0 [26.24 to 87.84]

4. Secondary Outcome: Duration of Response (DoR) as Assessed Based on RECIST v1.1
Description: The DoR was defined as the time, in days, from the first of the 2 assessments required for confirmed PR or CR to the time of the progressive disease (PD) or death due to underlying cancer. CR: Disappearance of all target or non-target lesions and normalization of tumor marker level. Any pathological lymph node (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. PD: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of the existing non-target lesions. The appearance of one or more new lesions was also considered progression.
Time Frame: From first dose of study drug until the date of first overall response of PD or date of death due to underlying cancer (maximum exposure: 638 days)
Population: RE Analysis Set: all participants with measurable disease at baseline who received study drug and had at least 1 post-baseline response assessment or discontinued treatment due to disease progression (including death due to disease progression) within 16 weeks of first dose of study drug. Per planned analysis, the efficacy data for Cohort F were collected and analyzed separately per tumor type. 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: days
Arm/Group | Cohort A: Endometrial Cancer CPI (PD-1/PD-L1) Naive | Cohort B: Head and Neck Squamous Cell Carcinoma | Cohort C: Cervical Carcinoma | Cohort E: TMB-H + MSS Solid Tumors | Cohort F: Rare Tumors (Uveal) | Cohort F: Rare Tumors (De-diff LPS) | Cohort F: Rare Tumors (UPS) | Cohort F: Rare Tumors (Other Sarcoma) | Cohort F: Rare Tumors (GCT) | Cohort G: Endometrial Cancer Post- CPI (PD-1/PD-L1 Treated) | Cohort H: Ovarian Cancer
Number analyzed (Participants) | 2 | 0 | 3 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1
days | 197.0 [57 to 337] |  | 183.0 [64 to 360] |  | 307.0 [92 to 522] | 464.0 [464 to 464] | 145.0 [145 to 145] |  |  |  | 442.0 [442 to 442]

5. Secondary Outcome: Duration of Stable Disease (DoSD) as Assessed Based on RECIST v1.1
Description: The DoSD was defined as the time, in days, from the first date of treatment until the first date at which PD was experienced or the participant died due to underlying cancer. PD: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of the existing non-target lesions. The appearance of one or more new lesions was also considered progression.
Time Frame: From first dose of study drug until the date of first overall response of PD or date of death due to underlying cancer (up to a maximum of 680 days)
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Cohort A: Endometrial Cancer CPI (PD-1/PD-L1) Naive | Cohort B: Head and Neck Squamous Cell Carcinoma | Cohort C: Cervical Carcinoma | Cohort E: TMB-H + MSS Solid Tumors | Cohort F: Rare Tumors (Uveal) | Cohort F: Rare Tumors (De-diff LPS) | Cohort F: Rare Tumors (UPS) | Cohort F: Rare Tumors (Other Sarcoma) | Cohort F: Rare Tumors (GCT) | Cohort G: Endometrial Cancer Post- CPI (PD-1/PD-L1 Treated) | Cohort H: Ovarian Cancer
Number analyzed (Participants) | 10 | 1 | 8 | 9 | 8 | 10 | 6 | 3 | 4 | 3 | 10
days | 81.5 [50 to 423] | 45.0 [45 to 45] | 120.0 [50 to 414] | 57.0 [45 to 140] | 109.5 [52 to 680] | 108.0 [36 to 568] | 55.5 [16 to 337] | 53.0 [52 to 60] | 57.5 [56 to 58] | 50.0 [50 to 58] | 70.0 [37 to 547]

6. Secondary Outcome: Serum Concentrations of Etigilimab
Time Frame: Pre-infusion and 15 minutes post-infusion on Cycle 1 Day 1 and Cycle 4 Day 43
Population: The pharmacokinetic (PK) analysis set included all participants with sufficient plasma concentration data to allow the characterization of the PK parameters. Per planned analysis, PK data were collected and analyzed combined for all arm groups. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms (μg)/milliliter (mL)
Groups:
- Etigilimab: Participants received etigilimab in combination with nivolumab every 2 weeks and continued treatment until protocol-defined discontinuation criteria were met.
Arm/Group | Etigilimab
Number analyzed (Participants) | 30
micrograms (μg)/milliliter (mL)
  Cycle 1 Day 1 (Pre-infusion) | NA (NA) — Sample below the limit of quantification (0.200 μg/mL).
  Cycle 1 Day 1 (15 minutes post-infusion): number analyzed (Participants) | 29
  Cycle 1 Day 1 (15 minutes post-infusion) | 262 (22)
  Cycle 4 Day 43 (Pre-infusion): number analyzed (Participants) | 25
  Cycle 4 Day 43 (Pre-infusion) | 20.1 (82)
  Cycle 4 Day 43 (15 minutes post-infusion): number analyzed (Participants) | 25
  Cycle 4 Day 43 (15 minutes post-infusion) | 273 (27)

7. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) to Etigilimab
Time Frame: as for outcome 2
Population: The immunogenicity analysis set included all participants with at least 1 evaluable post-treatment immunogenicity sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Endometrial Cancer CPI (PD-1/PD-L1) Naive | Cohort B: Head and Neck Squamous Cell Carcinoma | Cohort C: Cervical Carcinoma | Cohort E: TMB-H + MSS Solid Tumors | Cohort F: Rare Tumors (Sarcoma, Uveal Melanoma, Germ Cell) | Cohort G: Endometrial Cancer Post- CPI (PD-1/PD-L1 Treated) | Cohort H: Ovarian Cancer
Number analyzed (Participants) | 0 | 1 | 1 | 0 | 6 | 0 | 1
Participants |  | 0 | 0 |  | 0 |  | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 100 days after the last dose of study drug or the initiation of any subsequent cancer treatment, whichever occurs first (maximum exposure: 638 days)
Description: Safety Analysis Set included all participants who received any amount of study drug.
Arm/Group | Cohort A: Endometrial Cancer CPI (PD-1/PD-L1) Naive | Cohort B: Head and Neck Squamous Cell Carcinoma | Cohort C: Cervical Carcinoma | Cohort E: TMB-H + MSS Solid Tumors | Cohort F: Rare Tumors (Sarcoma, Uveal Melanoma, Germ Cell) | Cohort G: Endometrial Cancer Post- CPI (PD-1/PD-L1 Treated) | Cohort H: Ovarian Cancer
All-Cause Mortality (participants affected / at risk) | 2/11 | 1/1 | 2/8 | 5/9 | 14/33 | 2/4 | 5/10
Serious Adverse Events (participants affected / at risk) | 2/11 | 0/1 | 2/8 | 5/9 | 8/33 | 2/4 | 3/10
Other Adverse Events (participants affected / at risk) | 11/11 | 1/1 | 8/8 | 8/9 | 33/33 | 4/4 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Endometrial Cancer CPI (PD-1/PD-L1) Naive (N=11) | Cohort B: Head and Neck Squamous Cell Carcinoma (N=1) | Cohort C: Cervical Carcinoma (N=8) | Cohort E: TMB-H + MSS Solid Tumors (N=9) | Cohort F: Rare Tumors (Sarcoma, Uveal Melanoma, Germ Cell) (N=33) | Cohort G: Endometrial Cancer Post- CPI (PD-1/PD-L1 Treated) (N=4) | Cohort H: Ovarian Cancer (N=10)
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 2 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Abdominal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Immune-mediated gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malignant ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Endometrial Cancer CPI (PD-1/PD-L1) Naive (N=11) | Cohort B: Head and Neck Squamous Cell Carcinoma (N=1) | Cohort C: Cervical Carcinoma (N=8) | Cohort E: TMB-H + MSS Solid Tumors (N=9) | Cohort F: Rare Tumors (Sarcoma, Uveal Melanoma, Germ Cell) (N=33) | Cohort G: Endometrial Cancer Post- CPI (PD-1/PD-L1 Treated) (N=4) | Cohort H: Ovarian Cancer (N=10)
Nausea (Gastrointestinal disorders) | 4 | 0 | 3 | 3 | 6 | 0 | 5
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 4 | 3 | 5 | 0 | 3
Constipation (Gastrointestinal disorders) | 2 | 0 | 3 | 5 | 5 | 1 | 1
Vomiting (Gastrointestinal disorders) | 4 | 0 | 2 | 2 | 6 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2 | 3 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 0 | 1 | 1 | 11 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 1 | 5 | 0 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 5 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 0
Fatigue (General disorders) | 3 | 0 | 2 | 3 | 14 | 1 | 5
Oedema peripheral (General disorders) | 0 | 0 | 1 | 1 | 4 | 0 | 1
Chills (General disorders) | 2 | 0 | 0 | 1 | 3 | 0 | 0
Influenza like illness (General disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 2
Pyrexia (General disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1 | 4 | 2 | 3 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3 | 1 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 2 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 2 | 7 | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 1 | 4 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 1 | 7 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1 | 5 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 4 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 1 | 0 | 4 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 3 | 1 | 2 | 0 | 1
Weight decreased (Investigations) | 1 | 1 | 1 | 2 | 2 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 1 | 2 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 3 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 3 | 10 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0 | 5 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0 | 3 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 1 | 0 | 5 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All PIs must seek written permission from the sponsor before publication of any trial results.

DOCUMENTS (2):
  • Study Protocol (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/98/NCT04761198/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT04761198/SAP_001.pdf